CLINICAL TRIAL: NCT00684632
Title: A Phase III Clinical Study of KW-2246 for Breakthrough Pain in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2246-0702
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Pain, Cancer
Keywords: Pain, cancer
MeSH Terms: conditions — Cancer Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): KW-2246
  Interventions: Drug: KW-2246 (fentanyl citrate)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 2
Drug: KW-2246 (fentanyl citrate) — KW-2246 (fentanyl citrate)
  Arms: 1

SUMMARY:
This study is designed to determine whether KW-2246 is superior to placebo and not inferior to immediate-release morphine for the relief of breakthrough pain in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

At the time of obtaining written informed consent

* Provide written informed consent to participate in the study on a voluntary basis.
* Between the ages of 20 and 80 years (inclusive).
* Outpatients who live with a caregiver such as a family member, or inpatients.
* Regularly receiving one of the following opioid analgesics: sustained-release oral morphine, sustained-release oral oxycodone, and fentanyl transdermal patch.
* The daily dosage of the regular opioid analgesic regimen can be maintained constant from the baseline period through the end of the study as determined by the investigator.
* Require rescue medication at least 0.5 times (at least once every two days) but not more than three times per day on average as determined by the investigator.
* Performance Status (ECOG) of 3 or less at the time of giving written informed consent.Be able to receive diary training and have the ability to properly complete diaries as determined by the investigator.
* Have a life expectancy of at least three months as determined by the investigator.
* Be able to receive diary training and have the ability to properly complete diaries as determined by the investigator.

At the time of randomization

* The "regular opioid analgesic" being used at the time of giving written informed consent has been taken at a fixed dosage throughout the baseline period.
* The "immediate-release morphine" being used at the time of giving written informed consent (Opso® (morphine hydrochloride hydrate) oral solution, morphine hydrochloride (powder), or morphine hydrochloride tablets) has been taken at a fixed dosage of 5, 10, 15, or 20 mg/dose throughout the baseline period.
* Have received rescue medication at least 0.5 times but not more than three times per day on average during the baseline period.
* Have had a pain intensity of at least 3 cm as rated on a visual analog scale (VAS) immediately before each of two or more rescue doses of immediate-release morphine during the baseline period, and had a mean decrease of at least 1.8 cm and at least one-third in VAS-rated pain intensity at 30 minutes after dosing compared with the pre-dose value.
* Have received diary training and been able to properly complete diaries during the baseline period.

Exclusion Criteria:

At the time of obtaining written informed consent

* Intolerable adverse reactions (as defined in Attachment 3) to opioids.
* Serious respiratory dysfunction.
* Asthma.
* Serious bradyarrhythmia.
* Serious hepatic dysfunction.
* Serious renal dysfunction.
* Susceptibility to respiratory depression due to conditions such as increased intracranial pressure, head injury and brain tumor.
* Patients who have a history of clinically significant adverse reactions to the combination of opioid analgesics and any of the following drugs/substances, and who are currently receiving or expect to receive any of them during the study:

Central nervous system depressants (phenothiazines, benzodiazepines and barbiturates), inhalation anesthetics, monoamine oxidase inhibitors, tricyclic antidepressants, skeletal muscle relaxants, antihistamines, ritonavir, alcohol, itraconazole, amiodarone, clarithromycin, diltiazem, and fluvoxamine.

* History of convulsive seizures (except a single episode of infantile febrile convulsions).
* History of hypersensitivity to fentanyl.
* Current or past history of drug dependence or narcotic abuse.
* Pregnant or lactating women, possibly pregnant women, or women who are planning to become pregnant.
* Participation in any other clinical trial within 28 days prior to giving written informed consent.
* Prior exposure to KW-2246.
* Patients who are judged by the investigator/subinvestigator to be inappropriate for this study.

At the time of randomization

* Have experienced intolerable adverse reactions (as defined in Attachment 3) to opioids during the baseline period.
* Have received, during the baseline period, any morphine, oxycodone and fentanyl formulations other than the "regular opioid analgesic" being used at the time of giving written informed consent.
* Use of codeine, dihydrocodeine, opium, pethidine, buprenorphine, pentazocine, tramadol, butorphanol, and eptazocine within seven days prior to randomization (except codeine at daily dosages up to 60 mg and dihydrocodeine at daily dosages up to 30 mg for the treatment of cough).
* Interventions that may affect pain intensity rating, such as surgery, radiation therapy and nerve bThe daily dosages of systemically-acting adjuvant analgesics or drugs with analgesic activity have been modified during the baseline period.lock, within seven days prior to randomization.
* Use of narcotic antagonists within seven days prior to randomization.
* The daily dosages of systemically-acting adjuvant analgesics or drugs with analgesic activity have been modified during the baseline period.
* The daily dosages of locally-acting adjuvant analgesics or drugs with analgesic activity being used for the relief of cancer pain have been modified during the baseline period.
* The daily dosages of codeine (up to 60 mg/day) and dihydrocodeine (up to 30 mg/day) being used for the treatment of cough have been modified during the baseline period.
* Have the following results in the most recent laboratory tests conducted within seven days prior to randomization:

AST >5 times the upper limit of normal at each study site (ULN); ALT >5 times ULN; or Serum creatinine >1.5 times ULN.

* Dry mouth that affects sublingual administration (i.e., poor compliance during sublingual administration training with placebo).
* Subjects who are judged by the investigator/subinvestigator to be inappropriate for the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (20):
- Japan (20):
  - Nagoya, Aichi-ken
  - Katori-shi, Chiba
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Kōriyama, Fukushima
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Kasama, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Uji, Kyoto
  - Azumino, Nagano
  - Ibaraki, Osaka
  - Izumisano, Osaka
  - Mibu, Tochigi
  - Bunkyo-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Kumamoto
  - Okayama
  - Toyama
  - Wakayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimoyama N, Gomyo I, Teramoto O, Kojima K, Higuchi H, Yukitoshi N, Ohta E, Shimoyama M. Efficacy and safety of sublingual fentanyl orally disintegrating tablet at doses determined from oral morphine rescue doses in the treatment of breakthrough cancer pain. Jpn J Clin Oncol. 2015 Feb;45(2):189-96. doi: 10.1093/jjco/hyu182. Epub 2014 Nov 6. PMID 25378647